CLINICAL TRIAL: NCT02689700
Title: Examination of Diaplacental Transfer of IgG-antibodies Against Human Cytomegalovirus (HCMV) and Varicella-Zoster-Virus (VZV) at Premature and Mature Newborns
Brief Title: Diaplacental Transfer of Anti-HCMV- and Anti-VZV-immunoglobulin G (IgG) -Antibodies at Premature and Mature Newborns
Acronym: MoChi-HCMV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Horst Buxmann, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: 040713 FRA Mat Fet CMV Antib
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Materno-fetal Transfer of Anti-HCMV-IgG; Materno-fetal Transfer of Anti-VZV-IgG
Keywords: Human Cytomegalovirus; Varicella Zoster Virus; Materno-fetal antibody transfer; Pregnancy; Gestational age
MeSH Terms: conditions — Chickenpox | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Umbilical Cord blood; Blood from peripheral vene
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCMV antibody-transfer: Materno-fetal HCMV antibody-Transfer form 24-41 weeks of gestation
  Interventions: Other: Blood samples
- VZV antibody-transfer: Materno-fetal VZV antibody-Transfer form 24-41 weeks of gestation
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Taking blood form the umbilical cord (fetal circulation) and from the vein of the corresponding mother.

SUMMARY:
The aim of the study is to determine the total concentration of HCMV- and VZV-specific IgG-antibodies and the total concentration of neutralizing antibodies against HCMV in neonatal bloodstream depending on gestational age at birth.

DETAILED DESCRIPTION:
For data gathering the investigators measure the main concentration of specific HCMV-/VZV-IgG-antibodies and the concentration of neutralizing IgG-antibodies against HCMV and VZV in maternal blood and in fetal bloodstream. Then the investigators compare the data of mother and newborn. Therefore, the investigators use the following blood samples:

Mother: Venous blood sample taken at birth (+/- three days)

Newborn: Blood sample of umbilical cord (= fetal bloodstream) taken immediately after birth.

The investigators assign the data of each newborn (gestational age at birth) to the data of their respective mother for statistical evaluation. After finishing the study the investigators will destroy all residual blood.

ELIGIBILITY:
Inclusion Criteria:

* HCMV and/or VZV-seropositive pregnant woman who signed written informed consent form.

Exclusion Criteria:

* Newborns of underage mothers.
* Newborns whose mother did not sign the written informed consent.
* Pregnant women with a known hereditary or acquired immune deficiency

Ages: 1 Minute to 10 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Approximately 450 mother-child-pairs seropositive for HCMV and/or VZV
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
To measure the concentration of specific HCMV-/VZV-IgG-antibodies in fetal bloodstream depending on gestational age at birth. | Newborn: immediately after birth; Mother +/- 3 days at birth
  Measurement of HCMV and VZV-antibodies in the fetal and the maternal circulation

SECONDARY OUTCOMES:
Gauging the concentration of neutralizing IgG-antibodies against HCMV and VZV in fetal bloodstream depending on gestational age at birth. | Newborn: immediately after birth; Mother +/- 3 days at birth
  Measurement of neutralizing IgG-HCMV and VZV-antibodies in the fetal and the maternal circulation

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of the Johann Wolfgang-Goethe Univeristy, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hobbs JR, Davis JA. Serum gamma-G-globulin levels and gestational age in premature babies. Lancet. 1967 Apr 8;1(7493):757-9. doi: 10.1016/s0140-6736(67)91369-4. No abstract available. PMID 4164125
- [Result] Simister NE. Placental transport of immunoglobulin G. Vaccine. 2003 Jul 28;21(24):3365-9. doi: 10.1016/s0264-410x(03)00334-7. PMID 12850341
- [Result] Mussi-Pinhata MM, Pinto PC, Yamamoto AY, Berencsi K, de Souza CB, Andrea M, Duarte G, Jorge SM. Placental transfer of naturally acquired, maternal cytomegalovirus antibodies in term and preterm neonates. J Med Virol. 2003 Feb;69(2):232-9. doi: 10.1002/jmv.10271. PMID 12683413
- [Result] Linder N, Waintraub I, Smetana Z, Barzilai A, Lubin D, Mendelson E, Sirota L. Placental transfer and decay of varicella-zoster virus antibodies in preterm infants. J Pediatr. 2000 Jul;137(1):85-9. doi: 10.1067/mpd.2000.106902. PMID 10891827